CLINICAL TRIAL: NCT07281976
Title: An Open-label, Multicenter Phase Ib/II Clinical Study to Evaluate the Efficacy and Safety of LBL-024 Monotherapy or in Combination With Albumin-bound Paclitaxel in Patients With Recurrent or Metastatic Triple Negative Breast Cancer
Brief Title: A Trial of LBL-024 Monotherapy or Combination Drug in Patients With Triple Negative Breast Cancer
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Nanjing Leads Biolabs Co.,Ltd (Industry)
Collaborators: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LBL-024-CN005
Record Dates: First submitted 2025-12-02; First posted 2025-12-15 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-01

CONDITIONS: Triple Negative Breast Cancer
MeSH Terms: conditions — Triple Negative Breast Neoplasms | interventions — Injections; Albumin-Bound Paclitaxel; toripalimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LBL-024 + albumin-bound paclitaxel (Experimental): Experimental group：
  LBL-024 + albumin-bound paclitaxel.
  Intravenous infusion.
  Interventions: Drug: LBL-024 for Injection; Drug: albumin-bound Paclitaxel injection
- Toripalimab + albumin-bound paclitaxel/albumin-bound paclitaxel (Active Comparator): control group：
  Toripalimab + albumin-bound paclitaxel or albumin-bound paclitaxel.
  Intravenous infusion.
  Interventions: Drug: albumin-bound Paclitaxel injection; Drug: Toripalimab Injection

INTERVENTIONS:
Drug: LBL-024 for Injection — Intravenous infusion.
  Other Names: LBL-024
  Arms: LBL-024 + albumin-bound paclitaxel
Drug: albumin-bound Paclitaxel injection — Intravenous infusion.
  Other Names: albumin-bound Paclitaxel
Drug: Toripalimab Injection — Intravenous infusion.
  Other Names: Toripalimab
  Arms: Toripalimab + albumin-bound paclitaxel/albumin-bound paclitaxel

SUMMARY:
This trial is an open-label, multicenter phase Ib/II clinical study to evaluate the efficacy and safety of LBL-024 monotherapy or in combination with albumin-bound paclitaxel in patients with recurrent or metastatic triple negative breast cancer(TNBC).

DETAILED DESCRIPTION:
The trial was divided into two phases.

Stage I (Phase Ib):

Part A: Monotherapy Period:In the phase Ib Part A monotherapy period, a small number of TNBC patients were planned to be enrolled to receive LBL-024 monotherapy.The safety, tolerability, and preliminary efficacy of LBL-024 monotherapy in this population will be assessed by the sponsor and investigator in combination.

Part B: Combination Drug Safety Run-In Period:If the safety and tolerability are good and there is preliminary efficacy in Part A,The investigator discussed with the sponsor to decide whether to continue the study in Part B of Phase Ib.Part B is designed to enroll a small number of TNBC patients to receive LBL-024 combination therapy.

Stage II (Phase II) ： If the safety and tolerability are good and there is preliminary efficacy in the first stage,The investigator discusses with the sponsor to decide whether to continue the co-administration expansion study, continue to enroll TNBC patients, and using a randomized, open, positive control trial design.

This study will enroll up to 220 subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Agree to follow the trial treatment regimen, visit schedule, laboratory test, and other requirements of the protocol, and voluntarily enroll in the study and sign the written informed consent.
2. At the time of signing the informed consent form, the age was ≥ 18 years old.
3. The Eastern Cooperative Oncology Group's physical status scoring standard (ECOG) is 0~1.
4. The expected survival time is at least 12 weeks.
5. According to the evaluation of RECIST 1.1 （Response Evaluation Criteria in Solid Tumours），the subjects enrolled have at least one measurable lesion.
6. Females of childbearing age are willing to take highly effective contraceptive measures From the signing of the informed consent form to within 6 months after the last administration of the trial drug; Women of childbearing age must have a negative pregnancy test within 7 days before the first trial drug is administered.Male patients are willing to take highly effective contraceptive measures From the signing of the informed consent form to within 6 months after the last administration of the trial drug,and do not donate sperm during this period.

Exclusion Criteria:

1. Use of immunomodulatory drugs within 2 weeks prior to first dose of study drug.
2. Patients who received live vaccination within 4 weeks before the first dose of study drug or who are scheduled to receive live vaccination during the study treatment period and within 4 weeks after the last dose.
3. Patients with clinically uncontrolled pleural effusion, peritoneal effusion, or pericardial effusion.
4. Active infection within 2 weeks prior to first dose of study drug.
5. Active infectious disease.
6. Women with plans for pregnancy,Or women who are pregnant or breastfeeding.
7. Active hepatitis B or active hepatitis C.
8. History of mental illness (interfering with understanding or giving informed consent), drug abuse, alcoholism, or drug addiction.
9. The investigator believes that the subject has other conditions that may affect compliance or are not suitable for participating in this study.

   -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2026-01-27 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | From all subjects signed the informed consent form up to the completion of the follow-up period of drug withdrawal (28 days after drug withdrawal or before the start of new anti-tumor therapy)
  According to the evaluation criteria of RECIST V1.1 (solid tumour) ,Proportion of subjects achieving complete response (CR) or partial response (PR).It was used to evaluate the efficacy in Phase Ib.
Occurrence of adverse event (AE) and serious adverse event (SAE) | From all subjects signed the informed consent form up to the completion of the follow-up period of drug withdrawal (90 days after drug withdrawal or before the start of new anti-tumor therapy)
  Adverse event (AE) will be graded according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) 5.0.The safety profile of LBL-024 or LBL-024 Combination Administration will be assessed by monitoring the adverse event (AE) and serious adverse event (SAE) in Phase Ib study.
Progression-free Survival(PFS) | From all subjects signed the informed consent form up to the completion of the follow-up period of drug withdrawal (28 days after drug withdrawal or before the start of new anti-tumor therapy)
  According to the evaluation criteria of RECIST V1.1 (solid tumour),Time from randomisation to disease progression or death from any cause.It was used to evaluate Time of disease no-progression or Drug resistance in Phase II.

SECONDARY OUTCOMES:
Cmax | From all subjects signed the informed consent form up to the completion of the follow-up period of drug withdrawal (28 days after drug withdrawal or before the start of new anti-tumor therapy)
  Maximum drug concentration in plasma after administration.
Tmax | From all subjects signed the informed consent form up to the completion of the follow-up period of drug withdrawal (28 days after drug withdrawal or before the start of new anti-tumor therapy)
  After administration,Time to reach maximum drug concentration in plasma.
Immunogenicity | From all subjects signed the informed consent form up to the completion of the follow-up period of drug withdrawal (28 days after drug withdrawal or before the start of new anti-tumor therapy)
  The immunogenicity is evaluated by the incidence of anti-drug antibodies (ADA) and neutralizing antibodies (if applicable) in subjects.Immunogenicity refers to the performance that can elicit an immune response.
Disease Control Rate(DCR) | From all subjects signed the informed consent form up to the completion of the follow-up period of drug withdrawal (28 days after drug withdrawal or before the start of new anti-tumor therapy)
  Percentage of participants achieving CR, PR, iCR, iPR and stable disease (SD) after treatment.
Duration of Response(DOR) | From all subjects signed the informed consent form up to the completion of the follow-up period of drug withdrawal (28 days after drug withdrawal or before the start of new anti-tumor therapy)
  DOR is defined as the duration from earliest date of disease response (CR、PR 、iCR or iPR) until earliest date of disease progression or death from any cause(if occurring sooner than progression).

CONTACTS AND LOCATIONS:
Overall Officials: yongmei Yin, Principal Investigator — The First Affiliated Hospital with Nanjing Medical University
Locations (7):
- China (7):
  - Sun Yat-sen University Cancer Center, Guangzhou, Guangdong
  - Sun Yat-sen Memorial Hospital, Sun Yat-sen University, Guangzhou, Guangdong
  - Harbin Medical University Cancer Hospital, Harbin, Heilongjiang
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Jiangsu Province Hospital, Nanjing, Jiangsu
  - The first hospital of Jilin University, Changchun, Jilin
  - Liaoning Cancer Hospital, Shenyang, Liaoning

IPD SHARING:
Plan to Share IPD: No